CLINICAL TRIAL: NCT02926807
Title: Vascular Inflammation and Coronary Atherosclerosis Risks in Subjects With Atopic Dermatitis
Brief Title: Trial on Vascular Inflammation in Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Montreal Heart Institute (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: Inno-6043
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Atopic Dermatitis; Vascular Inflammation; Coronary Atherosclerosis
Keywords: Atopic Dermatitis; Vascular Inflammation; Coronary Atherosclerosis; Ascending aorta; Pet scan
MeSH Terms: conditions — Dermatitis, Atopic; Coronary Artery Disease | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atopic Dermatis Subjects: 30 subjects with atopic dermatitis
  Interventions: Other: FDG-PET Scan; Other: MDCT; Other: biopsy and blood collection
- Healthy Volunteers: 30 subjects without AD that matches for sex, age (± 2 years) and coronary artery disease risk factor with the AD subjects will be included as control case
  Interventions: Other: FDG-PET Scan; Other: MDCT; Other: biopsy and blood collection

INTERVENTIONS:
Other: FDG-PET Scan — a 18FDG-PET to quantify vascular inflammation
Other: MDCT — a MDCT to calculate the Agatston score
Other: biopsy and blood collection — biopsy and blood collection to assess biomarkers

SUMMARY:
A total of 30 subjects with moderate to severe atopic dermatitis. Thirty subjects without AD matched for sex, age and coronary artery disease risk factor with the AD subjects will also be included. All subjects will undergo the following imaging procedures: a 18FDG-PET to quantify vascular inflammation in the ascending aorta and carotids and a MDCT to calculate the Agatston score. Skin and blood biomarkers will also be assessed.

ELIGIBILITY:
Main inclusion Criteria:

* Men or women
* 18 years of age or older at time of consent.
* For AD subjects only: Confirmed clinical diagnosis of active AD according to Hanifin and Rajka criteria, BSA, EASI and IGA.
* For AD subjects only: Diagnosis of atopic dermatitis for at least 5 years.
* Women of childbearing potential is willing to use effective contraceptive method.
* Women of childbearing potential must have a negative urine pregnancy test.

Main exclusion Criteria:

* Has known cardiovascular arterial disease, a pacemaker, psoriasis, uncontrolled diabetes.
* Presence of an unstable co-morbidity that could have an effect on vascular inflammation.
* Heart rate restriction for patients with asthma or COPD.
* Use of any topical medication for atopic dermatitis on the site to be biopsied.
* Use of systemic treatments for atopic dermatitis.
* Use of phototherapy, tanning booth or other ultraviolet light sources.
* Use of biologics.
* Use of experimental medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 30 subjects with atopic dermatitis and 30 subjects without AD will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2017-01; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Target to background ratio (TBR) from the ascending aorta | 0 Days

SECONDARY OUTCOMES:
Target to background ratio (TBR) from the carotids | 0 Days
Agatston score | 0 Days

OTHER OUTCOMES:
Correlation between target to background ratio (TBR) and biomarkers, AD severity measurements (EASI, BSA, IGA and SCORAD), endothelial cell-derived micro particles. | 0 Days

CONTACTS AND LOCATIONS:
Overall Officials: Innovaderm Research clinical site, Principal Investigator — Innovaderm Research clinical site
Locations (1):
- Innovaderm Research Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No